CLINICAL TRIAL: NCT03637348
Title: Effect of TrueTear Use on Anterior Corneal Surface Imaging Quality
Brief Title: Effect of TrueTear Corneal Surface Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Price Vision Group (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-008
Record Dates: First submitted 2018-08-03; First posted 2018-08-20 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Cataract; Myopia
MeSH Terms: conditions — Cataract; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TrueTear (Other): Use of TrueTear device to stimulate tear production
  Interventions: Device: TrueTear

INTERVENTIONS:
Device: TrueTear — Ues of TrueTear neurostimulator

SUMMARY:
This study will evaluate the utility of TrueTear™ to improve anterior corneal surface imaging quality before cataract surgery, refractive lens exchange, or laser refractive surgery.

DETAILED DESCRIPTION:
Corneal imaging will be repeated before and after TrueTear use during a single patient visit. Image quality measures will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo routine imaging for cataract surgery, refractive lens exchange or laser refractive surgery

Exclusion Criteria:

* A cardiac pacemaker, implanted or wearable defibrillator, or other implanted metallic or electronic device (e.g. cochlear implant) in the head or neck
* Chronic or frequent nosebleeds, a bleeding disorder (e.g. hemophilia), or another condition that can lead to increased bleeding
* A known hypersensitivity (allergy) to the hydrogel material that comes into contact with the inside of the nose during use of the TrueTearTM device
* Pregnancy
* Presence of any ocular disease or condition which in the investigator's opinion would confound the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr., MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TrueTear: Use of TrueTear device to stimulate tear production
  TrueTear: Use of TrueTear neurostimulator
Period: Overall Study
Arm/Group | TrueTear
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TrueTear
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Surface Asymmetry Index (SAI) Assessed With Corneal Topography
Description: Surface asymmetry index (SAI) is an index that indicates an average value of the corneal power differences between the points spatially located at 180° from 128 equidistant meridians. A radially symmetrical surface has a value of zero, and this value increases as the degree of asymmetry is greater. Higher values are worse, but there is no set maximum value and no unit of measure.
Time Frame: Change from baseline SAI at 5-10 minutes after using the TrueTear device.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | TrueTear
Number analyzed (Participants) | 45
unitless | 0.21 (0.34)

2. Secondary Outcome: Surface Regularity Index (SRI) Assessed With Corneal Topography
Description: Surface Regularity index (SRI) is a local descriptor of surface regularity in a central 4.5 mm diameter area of the cornea. It correlates well with the value of visual acuity (p = 0.80, P <0.001), assuming the cornea is the only limiting factor for vision. A normal cornea presents SRI values below 0.56 (the SRI would be 0 in a perfectly regular cornea). SRI values increase with increasing irregularity of the corneal surface. Higher values are worse, but there is no set maximum value and no unit of measure.
Time Frame: Change from baseline SRI at 5-10 minutes after using the TrueTear device.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | TrueTear
Number analyzed (Participants) | 45
unitless | 0.1 (0.3)

ADVERSE EVENTS:
Time Frame: During the single study visit
Arm/Group | TrueTear
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03637348/Prot_SAP_000.pdf